CLINICAL TRIAL: NCT03453255
Title: Decitabine in Combination With Chidamide, Homoharringtonine and Ara-c (DCHA) as Postremission Therapy for Acute Myeloid Leukemia With t(8;21) :A Multicenter Prospective Study
Brief Title: DCHA as Postremission Therapy for AML With t(8;21)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Yu, MD. PH.D, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301-XYK-004
Record Dates: First submitted 2018-02-23; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Chemotherapy
Keywords: AML, chidamide, decitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- t(8;21)AML (Experimental): chemotherapy 5-Aza-2'-deoxycytidine IV 20mg/m2 d8-12 homoharringtonine IV 2mg d1-5 chidamide P.O. 30mg twice/W cytarabine IV 1000mg/m2(<60 year old) 500mg/m2(>60 year old) IV q12h d1,3,5
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — chidamide, decitabine, homoharringtonine, cytarabine
  Other Names: DCHA

SUMMARY:
Acute myelocytic leukemia ( AML) is a highly heterogeneous group of malignant hematopathy. Chromosomal translocation with t (8; 21) (q22; q22) , about 10 ~ 15% incidence in AML and 40% incidence in the AML-M2 type of leukemia, is a karyotype that is considered to have a good prognosis. The National Comprehensive Cancer Network (NCCN) guidelines recommend that high-dose Ara-c regimens may benefit for patients, but with 30 to 40% relapse and serious risks on myelosuppression, infection and bleeding in high-dose Ara-c consolidation chemotherapy and more than 70% recurrence rate with （tyrosine kinase）KIT mutation. So the exploration of a relatively safe and efficient consolidation therapy is one of the difficult problems to be solved in the treatment of mitigatory t (8; 21) AML.

DETAILED DESCRIPTION:
Treatment regimen

HA:

homoharringtonine 2mg IV d1-5 cytarabine( Ara-C) 1500mg/m2(<60 year old) ; 1000mg/m2(>60 year old) IV q12h

DCHA:

Decitabine 20mg/m2 d8-12 Chidamide 30mg twice/week P.O. for two weeks per cycle (four doses totally) cytarabine( Ara-C) 1500mg/m2(<60 year old) ; 1000mg/m2(>60 year old) IV q12h d1,3,5 homoharringtonine 2mg IV d10-14

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent provided.

  * The patients were diagnosed AML-M2 with t(8;21) (q22;q22) chromosomal changes and positive acute myeloid leukemia(AML1)-eight twenty one(ETO) fusion gene according to the 2008 World Health Organization (WHO) diagnostic criteria for malignant myeloid diseases.
  * Males or females aged ≥18 years, < 65 years.
  * Eastern Cooperative Oncology Group（ECOG） performance status 0-3.
  * Life expectancy ≥3 months.
  * The morphology was Complete remission (CR) or Cri after 2 cycles of anthracycline induced chemotherapy.
  * No serious disease with heart, lung, liver and kidney.
  * The ability to understand and be willing to sign the Informed Consent Form of the experiment.
  * Patient who can start the investigational therapy within 3-6 weeks after the complete resection
  * Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
  * Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
  * Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known allergic to prior treatment with drugs contained by the trial programme or with a chemical structure similar medicine.
* Pregnancy, breast-feeding women and childbearing age patients who do not want to take contraceptive measures.
* Active serious infection.
* Patients with extramedullary lesions.
* Patients who use drugs or drink alcohol for a long time to influence the evaluation of results.
* Patients with mental illness or other conditions are unable to obtain knowledge and consent, and can not cooperate with the requirements of the completion of the test treatment and examination steps.
* Patients with a history of the clinical significance of Q and T interval（QTc） prolongation (male > 450ms, female >470ms), ventricular tachycardia (VT), atrial fibrillation (AF), degree of heart block, muscle infarction (MI) within 1 years, congestive heart failure (CHF), with symptoms and drug therapy in patients with coronary heart disease.
* Patients with abnormal liver function (total bilirubin > 1.5 x ULN, ALT/AST > 2.5 x ULN, or liver invasion ALT/AST > 5x ULN ), renal function abnormality (serum creatinine > 1.5 x ULN).
* The researchers decided that patient was not appropriate to take part in the experiment.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  To evaluate the disease progression free survival of DCHA as postremission therapy for acute myeloid leukemia with t(8;21) . Progression free survival (PFS)- defined as the time from remission for the first time to the first documented disease progression.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival (OS)- defined as the length of time from trial treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, MD. Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT03453255/Prot_SAP_000.pdf